CLINICAL TRIAL: NCT04928560
Title: SMI and CEUS in the Diagnosis of Superficial Lymphadenopathy
Brief Title: Diagnosis of Superficial Lymphadenopathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-588
Record Dates: First submitted 2021-04-07; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-09

CONDITIONS: Lymphadenopathy; ULTRASOUND
MeSH Terms: conditions — Lymphadenopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- disease free survival: disease free survival
  Interventions: Diagnostic Test: SMI
- non-disease free survival: non-disease free survival
  Interventions: Diagnostic Test: SMI

INTERVENTIONS:
Diagnostic Test: SMI — ULTRASOUND
  Other Names: CEUS

SUMMARY:
The purpose of this study is to study the application of CEUS and SMI technology in superficial lymph node lesions (metastasis, lymphoma, inflammation, etc.), and to provide some diagnostic ideas for non-invasive diagnosis of lymph node lesions.

DETAILED DESCRIPTION:
CEUS and SMI technology were used to evaluated the superficial lymph node lesions (metastasis, lymphoma, inflammation, etc.), and to provide some diagnostic ideas for non-invasive diagnosis of lymph node lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 80 years old;
2. Patients with enlarged lymph nodes detected by ultrasound;
3. No contraindications such as hypersensitivity to contrast-enhanced ultrasound;
4. Voluntarily enrolled in this research project

Exclusion Criteria:

* The patient's position cannot be matched during ultrasound examination

  * Treatment history of lesion area: operation, radiotherapy, intervention, etc ③ Patients without informed consent ④ Lack of clinical data (no effective images such as two-dimensional ultrasound, color Doppler, contrast-enhanced ultrasound, micro blood flow imaging, or poor image quality, unable to analyze, unknown pathological results, etc.) ⑤ Lack of follow up information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with lymphadenopathy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
PATHOLOGY | up to 3 months
  BIOPSY/SURGERY

CONTACTS AND LOCATIONS:
Overall Officials: pintong Huang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- ZJU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided